CLINICAL TRIAL: NCT04086979
Title: Parents as Friendship Coaches for Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Parents as Friendship Coaches for Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Amori Yee Mikami, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 285413
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: ADHD
Keywords: friendship
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Coping Skills; Educational Status

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two interventions: Parental Friendship Coaching (PFC) or Coping with ADHD through Relationships and Education (CARE)
Who Masked: Outcomes Assessor
Masking Description: Some outcomes were observed by coders unaware of the participant's intervention condition. Other outcomes were reported by participants who were aware of their intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental Friendship Coaching (PFC) (Experimental)
  Interventions: Behavioral: Parental Friendship Coaching
- Coping with ADHD through Relationships and Education (CARE) (Active Comparator)
  Interventions: Behavioral: Coping with ADHD through Relationships and Education

INTERVENTIONS:
Behavioral: Parental Friendship Coaching — In this condition, therapists instructed parents in ways to coach their children to display better friendship behaviors using skills teaching, role play, active practice, and homework. This is a 10 week group intervention.
  Arms: Parental Friendship Coaching (PFC)
Behavioral: Coping with ADHD through Relationships and Education — In this condition, the therapist provided parents with psychoeducation about ADHD and friendship difficulties, and encouraged them to apply this information to their child and to support one another with tips about how to address these problems. This is a 10 week group intervention.
  Arms: Coping with ADHD through Relationships and Education (CARE)

SUMMARY:
Many children with Attention-Deficit/Hyperactivity Disorder (ADHD) have problems with making and keeping friends. The current study compared the efficacy of two 10-week behavioral interventions for improving the friendships of children with this disorder. Participants were children ages 6-11 with ADHD and their families, who were experiencing friendship problems. Outcome measures assessed friendship quality and friendship behaviors at baseline (pre-treatment), post-treatment, and 8-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children who meet diagnostic criteria for ADHD
* Children who are have peer relationship problems

Exclusion Criteria:

* Children with autism spectrum disorder, psychosis, or active suicidality (requires other interventions
* Children with intellectual disability (may not benefit from the interventions offered)
* Children who are not on a stable dose of medication (this treatment may affect outcome measures)
* Children who are receiving other behavioral treatment or treatment for social problems (these other treatments may affect outcome measures).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Friendship Quality - Questionnaires | change from baseline (pre-treatment) to post-treatment (approximately 4 months after baseline)
  Measures of positive and negative relationship quality with a friend, as reported by informants (adults, children) on the Friendship Quality Questionnaire
Change in Positive and Negative Friendship Quality - Questionnaires | change from baseline (pre-treatment) to follow-up (approximately 12 months after baseline, and 4 months after post-treatment)
  Measures of positive and negative relationship quality with a friend, as reported by informants (adults, children) on the Friendship Quality Questionnaire
Change in Positive and Negative Friendship Quality - Observations | change from baseline (pre-treatment) to post-treatment (approximately 4 months after baseline)
  Measures of positive and negative relationship quality with a friend, as observed in a lab-based interaction
Change in Positive and Negative Friendship Quality - Observations | change from baseline (pre-treatment) to follow-up (approximately 12 months after baseline, and 4 months after post-treatment)
  Measures of positive and negative relationship quality with a friend, as observed in a lab-based interaction

SECONDARY OUTCOMES:
Change in Positive and Negative Friendship Behaviors- Questionnaires | change from baseline (pre-treatment) to post-treatment (approximately 4 months after baseline)
  Measures of positive and negative behaviors with a friend, as reported by parents on the Quality of Play Questionnaire
Change in Positive and Negative Friendship Behaviors- Questionnaires | change from baseline (pre-treatment) to follow-up (approximately 12 months after baseline, and 4 months after post-treatment)
  Measures of positive and negative behaviors with a friend, as reported by parents on the Quality of Play Questionnaire
Change in Positive and Negative Friendship Behaviors- Questionnaires | change from baseline (pre-treatment) to post-treatment (approximately 4 months after baseline)
  Measures of positive and negative behaviors with a friend, as reported by parents and teachers on the Social Skills Informant System
Change in Positive and Negative Friendship Behaviors- Questionnaires | change from baseline (pre-treatment) to follow-up (approximately 12 months after baseline, and 4 months after post-treatment)
  Measures of positive and negative behaviors with a friend, as reported by parents and teachers on the Social Skills Informant System
Change in Positive and Negative Friendship Behaviors- Observations | change from baseline (pre-treatment) to post-treatment (approximately 4 months after baseline)
  Measures of positive and negative behaviors with a friend, as observed in a lab-based interaction
Change in Positive and Negative Friendship Behaviors- Observations | change from baseline (pre-treatment) to follow-up (approximately 12 months after baseline, and 4 months after post-treatment)
  Measures of positive and negative behaviors with a friend, as observed in a lab-based interaction

CONTACTS AND LOCATIONS:
Overall Officials: Amori Mikami, PhD, Principal Investigator — University of British Columbia; Sebastien Normand, PhD, Principal Investigator — Université du Québec en Outaouais

IPD SHARING:
Plan to Share IPD: No